CLINICAL TRIAL: NCT05334719
Title: A Non-interventional Observational Study of Effectiveness and Safety of Nivolumab Plus Chemotherapy for Untreated Advanced / Recurrent Gastric Cancer
Brief Title: A Study of the Effectiveness and Safety of Nivolumab Plus Chemotherapy in Participants With Untreated Advanced/Recurrent Gastric Cancer
Acronym: G-KNIGHT
Status: Active, not recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-6HP
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Stomach Neoplasms
Keywords: Nivolumab; Advanced or Recurrent; Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (1):
- Cohort 1: Participants with previously untreated advanced/recurrent gastric cancer (GC)

SUMMARY:
The purpose of this study is to assess the effectiveness, safety, and actual treatment status of first-line nivolumab plus chemotherapy in participants with untreated advanced / recurrent gastric cancer in a Japanese real-world setting.

DETAILED DESCRIPTION:
The Time Perspective for this observational study is defined as 'Retrospective and Prospective'.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced or recurrent gastric cancer
* Have initiated or are confirmed to receive nivolumab plus chemotherapy as the first-line therapy between the date of approval of nivolumab plus chemotherapy and December 31, 2022. For combination chemotherapy, SOX, CapeOX, or FOLFOX is acceptable
* Have signed a written informed consent form of their own free will after they have been given an adequate explanation and a full understanding of this study before enrolling in this study.

Exclusion Criteria:

* Treated with antineoplastic agents as first-line treatment for advanced or recurrent gastric cancer prior to the initiation of nivolumab plus chemotherapy (participants who have received prior perioperative chemotherapy and participants who have received prior bisphosphonates for osseous metastases may be enrolled)
* Confirmed to be positive for HER2
* Diagnosed with gastric cancer and have previously received investigational drugs with anti-tumor effects
* Initiated with nivolumab plus chemotherapy as the first-line treatment for advanced or recurrent gastric cancer at a site other than the study site and were later hospitalized at the study site.
* Judged by the investigators to be inappropriate for enrollment in this study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include participants who received nivolumab plus chemotherapy as first-line treatment for unresectable advanced or recurrent gastric cancer at least once between nivolumab plus chemotherapy approval and December 31, 2022.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2026-01-16 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 4 years
Objective response rate (ORR) | Up to approximately 4 years
Incidence of all immune-related adverse events (irAE) according to Common Terminology Criteria for Adverse Events (CTCAE) v5.0 | Up to approximately 4 years
Incidence of treatment-related adverse events (TRAE) that have led to treatment discontinuation | Up to approximately 4 years

SECONDARY OUTCOMES:
Overall survival (OS) | Up to approximately 4 years
Duration of response (DOR) | Up to approximately 4 years
Duration of treatment (DOT) | Up to approximately 4 years
Time to next treatment (TNT) | Up to approximately 4 years
Number of participants who have received subsequent therapy | Up to approximately 4 years
Incidence of Adverse Events (AEs) | Up to approximately 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Minato-ku, Tokyo, Japan

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm